CLINICAL TRIAL: NCT03552692
Title: A Phase II, Open Label, Multicenter Trial of Venetoclax (ABT-199/GDC-0199) as Single Agent in Patients With Relapsed/Refractory BCL-2 Positive Peripheral T Cell Lymphoma Not Otherwise Specified (PTCL-NOS), Angioimmunoblastic T-cell Lymphoma (AITL) and Other Nodal T-cell Lymphomas of T-follicular Helper Origin (TFH)
Brief Title: Use of Venetoclax as Single Agent in Patients With Relapsed/Refractory BCL-2 Positive Peripheral T Cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: efficacy lower than expected
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIL_VERT
Record Dates: First submitted 2018-05-10; First posted 2018-06-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: T-Cell Lymphoma Relapsed; T-Cell Lymphoma Refractory
Keywords: BCL-2 positive; PTCL-NOS; angioimmunoblastic T-cell lymphoma (AITL); T-follicular helper origin (TFH); Venetoclax; single agent
MeSH Terms: conditions — Immunoblastic Lymphadenopathy | interventions — venetoclax

STUDY DESIGN:
Intervention Model Description: Study design This is an open-label, multi-center, single arm phase II trial, with a two-stage design, to evaluate the activity and safety of ABT-199 single agent in patients with BCL-2 pos R/R PTCL-NOS, AITL, TFH.
  A pre-screening evaluation of immunohistochemical positivity of BCL-2 will be performed in the relapse biopsy, if available, or otherwise in the initial biopsy. BCL-2 evaluation will be centralized (FIL Laboratories). Only patients with a percentage of BCL-2 positive tumor cells ≥ 25% will be included onto the study. Patients will receive ABT-199 until disease progression, unacceptable toxicity, withdrawal of consent and/or the investigator determines that further therapy is not in the patient's best interest. The primary objective of the study is ORR which will be evaluated after 3 cycles of treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ARM1 - Venetoclax (ABT-199) (Experimental): Venetoclax (ABT-199) will be administered orally at the dose of 800 mg once daily.
  Response evaluation will be performed initially after 3 cycles from the beginning of treatment with ABT-199 and then every 3 cycles during the first 12 cycles, every 4 cycles from cycle 13 to 24; for those patients still on therapy after 24 cycles, the response evaluation, after this time, will be performed every 6 cycles.
  Interventions: Drug: Venetoclax

INTERVENTIONS:
Drug: Venetoclax — Venetoclax (ABT-199) will be administered orally (800 mg daily). Patients will receive ABT-199 until disease progression, unacceptable toxicity, withdrawal of consent and/or the investigator determines that further therapy is not in the patient's best interest.
  Tumor Lysis Syndrome (TLS) is an important identified risk for Venetoclax in oncology studies. Since there are no available data on the risk of TLS in PTCL, the risk of TLS development should be closely monitored during the study.
  to avoid TLS ABT-199 will be administered according the following ramp up: W eek 1 day 1: 20 mg W 1 day 2-3: 50 mg W 1 day 4-7: 100 mg W 2: 200 mg W 3: 400 mg W 4 and following: 800 mg
  Other Names: ABT-199/GDC-0199

SUMMARY:
The FIL_VERT study is a phase II, open label, multicenter clinical trial. The primary of objective of the Study is to evaluate the efficacy of Venetoclax ABT-199/GDC-0199) in terms of overall response rate (ORR) in patients with relapsed/refractory BCL-2 positive peripheral T cell lymphoma not otherwise specified (PTCL-NOS), angioimmunoblastic T-cell lymphoma (AITL) and other nodal T-cell lymphomas of T-follicular helper origin (TFH)

DETAILED DESCRIPTION:
This is an open-label, multi-center, single arm phase II trial, with a two-stage design, to evaluate the activity and safety of ABT-199 single agent in patients with BCL-2 pos R/R PTCL-NOS, AITL, TFH.

A pre-screening evaluation of immunohistochemical positivity of BCL-2 will be performed in the relapse biopsy, if available, or otherwise in the initial biopsy. BCL-2 evaluation will be centralized (FIL Laboratories). Only patients with a percentage of BCL-2 positive tumor cells ≥ 25% will be included onto the study. Patients will receive ABT-199 until disease progression, unacceptable toxicity, withdrawal of consent and/or the investigator determines that further therapy is not in the patient's best interest. The primary objective of the study is ORR which will be evaluated after 3 cycles of treatment.

ABT-199 will be administered orally at the dose of 800 mg once daily. Patients will receive ABT-199 until disease progression, unacceptable toxicity, withdrawal of consent and/or the investigator determines that further therapy is not in the patient's best interest (e.g., due to non-compliance, toxicity...) Response evaluation will be performed initially after 3 cycles from the beginning of treatment with ABT-199 (Response Assessment 1) and then every 3 cycles during the first 12 cycles, every 4 cycles from cycle 13 to 24; for those patients still on therapy after 24 cycles, the response evaluation, after this time, will be performed every 6 cycles.

Response will be evaluated according to the Lugano 2014 classification.

TLS is an important identified risk for ABT-199 in oncology studies, especially in CLL. Since there are no available data on the risk of TLS in PTCL, the risk of TLS development should be closely monitored during the study.

TLS prophylaxis includes:

1. ABT-199 will be administered according the following ramp up:

   * week 1 day 1: 20 mg
   * week 1 day 2-3: 50 mg
   * week 1 day 4-7: 100 mg
   * week 2: 200 mg
   * week 3: 400 mg
   * week 4 and following: 800 mg
2. Hospitalization and monitoring of the subject should occur for a minimum of 72 hours after the initial dose. Discharge of the subject is dependent upon review of chemistry labs 72 hours after the first dose of ABT-199
3. IV hydration (150 cc/hr, as tolerable) must be started upon admission and continued during hospitalization at least for 72 hours after the initial dose of ABT-199. Urine output must be monitored
4. Allopurinol 300 mg daily to be initiated 3 days before treatment and continued for up to 5 weeks based on the ongoing risk of TLS development. Subjects allergic to allopurinol must use another anti-hypeuricemic drug. Consider use of rasburicase if subjects baseline uric acid level is elevated
5. The investigator decision to proceed with ABT-199 treatment initiation and subsequent ramp up will be after having evaluated the normal value of the following biochemistry (potassium, uric acid, phosphorus, calcium and creatinine).

Biohemistry labs (potassium, uric acid, phosphorus, calcium and creatinine) must be performed as follow:

* week 1 (ABT-199 dose from 20 to 100 mg/daily): at timepoints 0 (pre-dose, within 4 hours from ABT-199 administration), 6-8, 24, 48, 72, 96 hours after the first dose of ABT-199. Day 2 dose should not be administered until the 24 hours post-dose labs are reviewed by the investigator;
* week 2 (ABT-199 dose 200 mg/daily): at timepoints 0 (pre-dose, with-in 4 hours from ABT-199 administration), 6-8, 24 hours after. Day 2 dose should not be administered until the 24 hours post-dose labs are reviewed by the investigator;
* week 3 (ABT-199 dose 400 mg/daily): at timepoints 0 (pre-dose, with-in 4 hours from ABT-199 administration), 6-8, 24 hours after. Day 2 dose should not be administered until the 24 hours post-dose labs are reviewed by the investigator;
* week 4 (ABT-199 dose 800 mg/daily): at timepoints 0 (pre-dose, with-in 4 hours from ABT-199 administration), 6-8, 24 hours after. Day 2 dose should not be administered until the 24 hours post-dose labs are reviewed by the investigator Nephrology (or other acute dialysis service) must be consulted/contacted on admission (per institutional standards to ensure emergency dialysis is available).

The efficacy interim analysis will be performed after enrollment of 18 patients. It is to be planned a stop in recruitment of at least 3 months to have the results of response assessment. The primary efficacy analysis will consist of an estimate of ORR on the efficacy population after the first 3 cycles of therapy, with 90% confidence intervals (according to 1-sided alpha error of 0.05). To proceed to the second stage, the minimum number of patients with an ORR is 3/18.

ELIGIBILITY:
Inclusion criteria:

* Histologically documented diagnosis of BCL-2 positive PTCL-NOS, AITL, TFH as defined in the 2016 edition of the World Health Organization (WHO) classification. Only patients with percentage of BCL-2 positive tu-mor cells ≥ 25% in the relapse biopsy, if available, or otherwise in the ini-tial biopsy, will be included onto the study;
* Age ≥ 18 years
* Relapsed or refractory to at least one previous standard line of treatment
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 2
* At least one site of measurable nodal or extranodal disease at baseline ≥ 2.0 cm in the longest transverse diameter as determined by CT scan (MRI is allowed only if CT scan cannot be performed). Note: Patients with only bone marrow involvement are eligible
* Adequate hematological counts defined as follows:
* Absolute Neutrophil count (ANC) > 1.0 x 10^9/L unless due to bone marrow involvement by lymphoma
* Platelet count ≥ 50.000/mm^3 unless due to bone marrow involvement by lymphoma
* Adequate renal function defined as follows:
* Creatinine clearance ≥ 30 mL/min
* Adequate hepatic function per local laboratory reference range as follows:
* Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3.0 x ULN
* Bilirubin ≤1.5 x ULN (unless bilirubin rise is due to Gilbert's syn-drome or of non-hepatic origin)
* Subject understands and voluntarily signs an informed consent form ap-proved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to the initiation of any screening or study-specific pro-cedures
* Subject must be able to adhere to the study visit schedule and other pro-tocol requirements
* Subject must be able to swallow capsules or tablets
* Life expectancy ≥ 3 months
* Women must be:
* postmenopausal for at least 1 year (must not have had a natural menses for at least 12 months)
* surgically sterile (have had a hysterectomy or bilateral oophorectomy, tubal ligation, or otherwise be incapable of pregnancy),
* completely abstinent (periodic abstinence from intercourse is not per-mitted) or if sexually active, be practicing a highly effective method of birth control (e.g., prescription oral contraceptives, contraceptive injec-tions, contraceptive patch, intrauterine device, double barrier method (e.g.: condoms, diaphragm, or cervical cap, with spermicidal foam, cream, or gel, male partner sterilization) as local regulations permit, be-fore entry, and must agree to continue to use the same method of con-traception throughout the study. They must also be prepared to contin-ue birth control measures for at least 1 month after terminating treat-ment.
* women of childbearing potential must have a negative pregnancy test at screening
* Men must agree to use an acceptable method of contraception (fort themselves or female partners as listed above) for the duration of the study. Men must agree to use a double barrier method of birth control and to not donate sperm during the study and for 1 month after receiving the last dose of study drug.

Male even if surgically sterilized (i.e., status postvasectomy) must agree to 1 of the following:

* practice effective barrier contraception during the entire study treatment period and through 1 months after the last dose of study drug, or
* agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods for the female part-ner] and withdrawal are not acceptable methods of contraception)

Exclusion criteria

* Histological diagnosis different from BCL-2 positive PTCL-NOS, AITL, and TFH
* Allogeneic or autologous stem cell transplant within 6 months prior to the informed consent signature
* Treatment with any of the following within 7 days prior to the first dose of study drug:
* steroid therapy for anti-neoplastic intent
* moderate or strong cytochrome P450 3A (CYP3A) inhibitors (see Ap-pendix C for examples)
* moderate or strong CYP3A inducers (see Appendix C for examples)
* Subject has received any anti-cancer therapy including chemotherapy, immunotherapy, radiotherapy, investigational therapy, including targeted small molecule agents within 14 days prior to the first dose of study drug
* History of CNS involvement by lymphoma
* Administration or consumption of any of the following within 3 days prior to the first dose of study drug:
* grapefruit or grapefruit products
* Seville oranges (including marmalade containing Seville oranges)
* star fruit
* Previous treatment with a BCL-2 family protein inhibitor
* Subject is known to be positive for HIV (HIV testing is not required)
* Cardiovascular disease (NYHA class ≥2)
* Creatinine Clearance < 30 mL/min
* Significant history of neurologic, psychiatric, endocrinologic, metabolic, immunologic, or hepatic disease that would preclude participation in the study or compromise ability to give informed consent.
* Any history of other active malignancies within 3 years prior to study en-try, with the exception of adequately treated in situ carcinoma of the cer-vix uterine, basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin, previous malignancy confined and surgically re-sected with curative intent.
* Subject who has malabsorption syndrome or other condition which pre-cludes enteral route of administration.
* Evidence of other clinically significant uncontrolled condition(s) including, but not limited to uncontrolled and/or active systemic infection (viral, bac-terial or fungal)
* Active HBV positive hepatitis
* The following categories of patients HBV positive but with non evidence of active hepatitis may be considered for the study:
* HBsAg positive with HBV DNA < 2000 UI/ml (inactive carriers); HBV DNA > 2000 UI/ml is criteria of exclusion
* HBsAg negative but HBsAb positive
* HBsAg negative but HBcAb positive
* Patients HBsAg positive with HBV DNA < 2000 UI/ml and HBsAg nega-tive but HBcAb positive will be eligible for the study only if they accept to receive prophylactic Lamivudine 100 mg/daily for all the period of treatment and at least for 12 months after the end of therapy. Treatment with ABT-199 should be stopped in case of hepatitis reactivation.
* Active HCV positive hepatitis
* If female, the patient is pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | After the first 3 cycles (each cycle is 28 days)
  Overall response rate (ORR) will be defined as the proportion of patient in CR or PR according to Re-sponse Criteria (Lugano 2014) after the first 3 cycles. Efficacy will be assessed after the first 3 cycles or, in case of discontinuation, at the EoT visit. Patients without response assessment (due to whatever reason) will be considered as non-responders.

SECONDARY OUTCOMES:
Complete remission (CR) | After the first 3 cycles (each cycle is 28 days)
  CR rate will be defined according to Lugano criteria21 after the first 3 cycles and at each restaging. The best overall response will be defined as the best response between the date of begin-ning of therapy and the last restaging. Patients without response assessment (due to whatever rea-son) will be considered as non-responders
Partial response (PR) | After the first 3 cycles (each cycle is 28 days)
  PR rate will be defined according to Lugano criteria21 after the first 3 cycles and at each restaging. The best overall response will be defined as the best response between the date of begin-ning of therapy and the last restaging. Patients without response assessment (due to whatever rea-son) will be considered as non-responders.
Stable Desease (SD) | After the first 3 cycles (each cycle is 28 days)
  SD rate will be defined according to Lugano criteria21 after the first 3 cycles and at each restaging. The best overall response will be defined as the best response between the date of begin-ning of therapy and the last restaging. Patients without response assessment (due to whatever rea-son) will be considered as non-responders.
Time To Response (TTR) | 1 year from the date of the first dose
  TTR will be defined for all patients who achieved a response (CR or PR) and is measured from the date of beginning of therapy until the date of response. Patients in relapse or progression will be cen-sored at their last assessment date. Patients death due to any cause will be consider censored or competing event according to different analysis plan
Duration of Remission (DoR) | 6 months from the first 3 cycles (each cycle is 28 days)
  DoR will be defined for all patients who achieved a response (CR or PR) and it is measured from the time of response until the date of progression or relapse. Patients without relapse or progression will be censored at their last assessment date; Patients death due to any cause will be consider censored or competing event according to different analysis plan;
Progression free Sruvival (PFS) | 1 year from the date of the first dose
  PFS will be defined as the time from beginning of therapy until lymphoma relapse or progression or death as a result of any cause; responding patients and patients who are lost to follow up will be cen-sored at their last assessment date;
Overall Survival (OS) | 1 year from the date of the first dose
  OS will be defined as the time from beginning of therapy until death as a result of any cause; patients alive will be censored at their last assessment date;
Duration of treatment (DoT) | 1 year from the date of the first dose
  Duration of treatment (DoT) will be defined as the time from beginning of therapy until ABT-199 dis-continuation due to any reason;
Toxicity - Incidence of Adverse Events | Through study completion, up to 30 months
  Safety of ABT-199 in terms of relevant toxicity and of overall toxicity (as acute and long-term toxicity). Toxicity will be classified according to definitions of Common Terminology Criteria for Adverse Event version 4.03 (CTCAE) commencing during and up to 24 hours after the first drug infusion and at any time during therapy and follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Zaja, MD, Principal Investigator — Azienda Sanitaria Universitaria Integrata di Trieste
Locations (13):
- Italy (13):
  - Centro Riferimento Oncologico - S.O.C. Oncologia Medica A, Aviano
  - Policlinico S.Orsola-Malpighi - Istituto di Ematologia "Seragnoli", Bologna
  - ASST Spedali Civili di Brescia - Ematologia, Brescia
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano - Ematologia, Milan
  - Istituto Scientifico San Raffaele - Unità Linfomi - Dipartimento Oncoematologia, Milan
  - AOU Maggiore della Carità di Novara - SCDU Ematologia, Novara
  - IRCCS Policlinico S. Matteo di Pavia - Div. di Ematologia, Pavia
  - Ospedale delle Croci - Ematologia, Ravenna
  - Azienda Unità Sanitaria Locale-IRCCS - Arcispedale Santa Maria Nuova - Ematologia, Reggio Emilia
  - Azienda sanitaria-universitaria integrata Trieste-SC Ematologia, Trieste
  - Azienda Sanitaria Universitaria Integrata di Udine (A.S.U.I. Udine) - SOC Clinica Ematologica, Udine
  - Ospedale di Circolo - U.O.C Ematologia, Varese
  - ULSS 8 Berica - Ospedale S. Bortolo - Ematologia, Vicenza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ballotta L, Zinzani PL, Pileri S, Bruna R, Tani M, Casadei B, Tabanelli V, Volpetti S, Luminari S, Corradini P, Lucchini E, Tisi MC, Merli M, Re A, Varettoni M, Pesce EA, Zaja F. Venetoclax Shows Low Therapeutic Activity in BCL2-Positive Relapsed/Refractory Peripheral T-Cell Lymphoma: A Phase 2 Study of the Fondazione Italiana Linfomi. Front Oncol. 2021 Dec 6;11:789891. doi: 10.3389/fonc.2021.789891. eCollection 2021. PMID 34938664